CLINICAL TRIAL: NCT06597643
Title: The Effect of Adding Deep Friction Massage to Eccentric Training Exercises in Lateral Epicondylitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Abdelkader Abdallah, Director, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005344
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lateral Epicondylitis (tennis Elbow)
Keywords: Lateral Epicondylitis; Eccentric Training; Deep Friction Massage (DFM; Wrist Extensor Strength
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: statistician will be blind to the details of allocation and intervention in each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Twenty-one patients will be assigned to group A, who will receive eccentric exercise program in addition to sham massage in the form of skin rubbing for patient blinding. for a total of 12 treatment sessions (3 sessions per week) for 4 weeks 3 sets of 15 repetitions, it takes 5 seconds to complete each repetition and between each set there is 30 seconds of rest
  Interventions: Other: Eccentric Training
- Experimental Group (Experimental): Twenty-one patients will be assigned to group B who will receive the same exercises as in control group (eccentric training exercises) in addition to deep friction massage (DFM) for a total of 12 treatment sessions (3 sessions per week) for 4 weeks. Before starting the exercises DFM will be performed. The patient will sit on a chair while holding a pillow. DFM will be performed in perpendicular direction to the Extensor carpi radialis brevis tendon the site of the application will be on the upper attachment of the common extensor origin (palpated one cm distal to the lateral epicondyle of the humerus) for 5 minutes. Using the thumb, Firm pressure will be applied to compress the extensor tendons, their origins, and the musculotendinous junctions between the underlying bone and the fingertips. This pressure will be maintained while the therapist applies DFM in the direction of their fingers,
  Interventions: Other: Eccentric Training; Other: Deep Friction Massage

INTERVENTIONS:
Other: Eccentric Training — Exercise 1: Eccentric Wrist Extension with Dumbbell
  Position: Seated, elbow extended, wrist maximally extended.
  Action:
  Lower: Slowly flex the wrist for 30 seconds. Return: Use the opposite hand to bring wrist back to extension. Load: Increase weight based on 10 Repetition Maximum (10RM). Exercise 2: Eccentric Wrist Extension with Twist-Bar
  Position: Hold Flex Bar with involved hand in extension.
  Action:
  Twist: Rotate the bar with the non-involved hand while keeping the involved wrist extended.
  Untwist: Allow the wrist to flex slowly. Exercise 3: Eccentric Supination with Elastic Band
  Position: Anchor band, elbow flexed to 90°.
  Action:
  Supinate: Rotate forearm with palm up. Flex: Slowly rotate to palm down, then return
Other: Deep Friction Massage — The patient will sit on a chair while holding a pillow. DFM will be performed in perpendicular direction to the Extensor carpi radialis brevis tendon the site of the application will be on the upper attachment of the common extensor origin (palpated one cm distal to the lateral epicondyle of the humerus) for 5 minutes. Using the thumb, Firm pressure will be applied to compress the extensor tendons, their origins, and the musculotendinous junctions between the underlying bone and the fingertips. This pressure will be maintained while the therapist applies DFM in the direction of their fingers,
  Arms: Experimental Group

SUMMARY:
Background: Lateral epicondylitis (LE) often benefits from eccentric training exercises, but combining them with deep friction massage (DFM) might enhance outcomes.

Objective: To evaluate if adding DFM to eccentric training improves pain, function, wrist extensor strength, and hand grip strength more than eccentric training alone.

Design: A triple-blinded, randomized controlled trial involving 46 participants aged 16-30 with unilateral LE. Participants will be randomly assigned to receive either eccentric training plus sham massage (Control Group) or eccentric training plus DFM (Experimental Group) over 4 weeks.

Methods: Outcomes will be measured using the Visual Analogue Scale (VAS) for pain, the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire for function, a hand-held dynamometer for wrist extensor strength, and a grip dynamometer for hand grip strength.

Blinding: The study is triple-blinded-assessors, statisticians, and participants are unaware of group allocations.

Significance: This study aims to determine if DFM enhances the effectiveness of eccentric training in LE rehabilitation, potentially leading to improved treatment protocols.

DETAILED DESCRIPTION:
Background: Lateral epicondylitis (LE), also known as tennis elbow, is an overuse injury of the elbow characterized by pain and functional impairment in the lateral aspect of the elbow. Traditional management strategies often include eccentric training exercises aimed at improving muscle strength and reducing pain. However, the addition of deep friction massage (DFM) to such a regimen might offer additional benefits.

Objective: This study aims to evaluate the impact of combining deep friction massage with eccentric training exercises on pain, functional ability, wrist extensor strength, and hand grip strength in patients with unilateral lateral epicondylitis.

Design: A triple-blinded randomized controlled trial (RCT) will be carried out at the outpatient physical therapy clinic of Pharos University in Alexandria, Egypt. The trial is designed to assess whether the integration of DFM with eccentric training offers superior outcomes compared to eccentric training alone.

Participants: The study will involve 46 patients aged 16 to 30 years, diagnosed with unilateral lateral epicondylitis. Participants will be randomly assigned to one of two groups: Group A (Control) and Group B (Experimental). Inclusion criteria include unilateral elbow pain, a BMI between 18.5 and 29.9, and chronic LE not treated with physical therapy in the past six months. Exclusion criteria include significant injuries or diseases affecting the shoulder, elbow, or wrist, recent local steroid injections, cervical radiculopathy, and neurological impairments.

Interventions:

Control Group (Group A): Participants will receive eccentric training exercises and sham massage. The eccentric training regimen includes three exercises: eccentric wrist extension with dumbbells, eccentric wrist extension with a twist-bar, and eccentric supination with an elastic band. Sham massage will be used to maintain blinding.

Experimental Group (Group B): Participants will receive the same eccentric training exercises as Group A, plus deep friction massage (DFM). DFM will be applied to the extensor carpi radialis brevis tendon at the site of the common extensor origin, with firm pressure applied perpendicular to the tendon for 5 minutes before each exercise session.

Outcome Measures:

Pain: Assessed using the Visual Analogue Scale (VAS), which allows patients to rate pain intensity on a 100 mm line ranging from "no pain" to "worst pain." Function: Evaluated using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, which includes 30 items measuring both function and symptoms in upper limb activities. Scores range from 0 (no disability) to 100 (severe disability).

Wrist Extensor Strength: Measured with a hand-held dynamometer, quantifying the maximum isometric strength of wrist extensors.

Hand Grip Strength: Assessed using a Jamar grip dynamometer, recording the maximum grip strength in kilograms.

Blinding and Randomization: The study will use a triple-blinding approach. Research assistants conducting assessments will be blinded to group allocations, as will the statisticians analyzing the data. Participants will also be unaware of their group assignment. Randomization will be achieved using an online random number generator to ensure unbiased group assignment.

Significance: This study seeks to determine if combining deep friction massage with eccentric training provides additional benefits over eccentric training alone in terms of pain reduction, functional improvement, and strength enhancement in patients with lateral epicondylitis. The results could inform more effective rehabilitation strategies for this common condition.

ELIGIBILITY:
Inclusion Criteria:

* Both gender male and female
* Age from 16 to 30
* Unilateral elbow pain
* Body mass index ranges from 18.5 to 29.9
* Non athletic patient
* Chronic LE don't receive PT for 6 months

Exclusion Criteria:

* Any injury or disease around the shoulder, elbow and wrist on the affected side
* Any b local intervention such as injection of steroids 6 month prior to the intervention
* Cervical radiculopathy
* History of fracture of radius, ulna and humerus with resultant deformity of the affected extremity
* Neurological impairments

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  is used to measure the pain which is represented from (0) grade to (10) grade, with zero means no pain and ten means intolerable pain, The subjects were asked to indicate the level of pain by placing a dash at the appropriate level on the 10 cm horizontal line

SECONDARY OUTCOMES:
-Disability of the Arm, Shoulder and Hand questionnaire Arabic version | 4 weeks
  It is a 30-item; self-report questionnaire designed to assess the patient's health status. The items indicate the degree of difficulty in performing different physical activities (21 items), the severity of each of the symptoms of pain, activity-related pain, tingling, weakness and stiffness (5 items) and the impact of the problem on social, work, sleep and self-image (4 items). Each item has 5 response options. Scores range from 0 (no disability) to 100 (most severe disability)
Hand-held Dynamometer | 4 weeks
  for measuring wrist extensor strength, it is a sensitive, objective and affordable device
-Jamar grip dynamometer | 4 weeks
  for measuring hand grip strength, it is an accurate and quantifiable assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Enas Fawzy yousef, Phd, Study Chair — Cairo University; Mai Mohamed Abdelkader, PhD, Study Director — Pharos university in alexanderia; sherif Hamdy Zawam, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vieira CS, Pack A, Roberts K, Davis AR. A pilot study of levonorgestrel concentrations and bleeding patterns in women with epilepsy using a levonorgestrel IUD and treated with antiepileptic drugs. Contraception. 2019 Apr;99(4):251-255. doi: 10.1016/j.contraception.2018.11.018. Epub 2018 Dec 4. PMID 30529085
- [Background] Libby AM, Pace W, Bryan C, Anderson HO, Ellis SL, Allen RR, Brandt E, Huebschmann AG, West D, Valuck RJ. Comparative effectiveness research in DARTNet primary care practices: point of care data collection on hypoglycemia and over-the-counter and herbal use among patients diagnosed with diabetes. Med Care. 2010 Jun;48(6 Suppl):S39-44. doi: 10.1097/MLR.0b013e3181ddc7b0. PMID 20473193
- [Background] Pietrini V, Pavesi G, Andreetta F. Miller Fisher syndrome with positivity of anti-GAD antibodies. Clin Neurol Neurosurg. 2013 Nov;115(11):2399-400. doi: 10.1016/j.clineuro.2013.09.002. Epub 2013 Sep 16. No abstract available. PMID 24094904
- See also: Lateral epicondylitis: a review of pathology and management. The bone & joint journal — https://pubmed.ncbi.nlm.nih.gov/24094904/
- See also: Lateral Elbow Tendinopathy: Development of a Pathophysiology-Based Treatment Algorithm — https://pubmed.ncbi.nlm.nih.gov/27833925/